CLINICAL TRIAL: NCT00837005
Title: Prognostic Value of High Dose Dobutamine Stress Magnetic Resonance in Patients With Ischemic Heart Disease. Assessment of Myocardial Perfusion and Wall Motion.
Brief Title: Prognostic Value of High Dose Dobutamine Stress Magnetic Resonance Imaging
Acronym: DS-Prognosis
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, G. Korosoglou, Prof. Dr., Heidelberg University
Other Study IDs: DOBU-STRESS01
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: dobutamine stress; inducible ischemia; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with suspected CAD
- 2: Patients with known CAD and suspected ischemia.

SUMMARY:
High-dose dobutamine/atropine stress cardiac magnetic resonance imaging (DS-MRI) has been incorporated in daily clinical practice for the detection of ischemic heart disease.

Thus, wall motion abnormalities (WMA) during stress, precede the development of ST-segment depression on ECG and of anginal symptoms and aid in the detection of anatomically significant coronary artery disease (CAD).

DS-MRI offers the possibility to integrate myocardial perfusion and wall motion analysis in a single examination. In this regard, recent data suggest that the assessment of myocardial wall motion and perfusion during a single session may enhance the sensitivity of the technique for the diagnosis of CAD.

However, to date limited data is available on the prognostic value of high-dose DS-MRI in large patient cohorts, treated according to current guidelines.

Assessment of long-term outcome of DS-MRI is important because this test may identify both high-risk patients, who would benefit from invasive diagnostic and therapy, and lower-risk patients in whom additional procedures and intensive medical follow-up are not required.

In the present study we aim to determine the value of wall motion and perfusion assessment during high-dose dobutamine/atropine MRI in predicting cardiac events.

In addition, the incremental value of the MR-stress testing results was assessed (inducible wall motion, perfusion abnormalities and the combination of both) after the consideration of traditional clinical risk factors and baseline ejection fraction.

DETAILED DESCRIPTION:
Background: High-dose dobutamine stress cardiac magnetic resonance imaging (DS-MRI) is incorporated in daily clinical practice for the detection of coronary artery disease (CAD). Purpose: To determine the value of wall motion and perfusion assessment during DS-MRI for the prediction of cardiac events in a large patient cohort.

Methods:

Cardiovascular MR-Examination. Patients are examined in a clinical 1.5-T whole-body MR-scanner Achieva system (Philips Medical Systems, Best, The Netherlands) using a 5-element cardiac phased-array receiver coil. Cardiovascular MR-images were acquired at rest and during a standardized high-dose dobutamine/atropine protocol involving short breath holds, and using a vector electrocardiogram for R-wave triggering11. Electrocardiographic rhythm and symptoms were monitored continuously, and blood pressure was measured every 3 minutes.

Follow-up Data. Personnel unaware of the stress testing results contacts each subject or an immediate family member and the date of this contact was used for calculating the follow-up time duration. Outcome data iscollected from a standardized questionnaire and determined from patient interviews at the outpatient clinic or by telephone interviews. Reported clinical events are confirmed by review of the corresponding medical records in our electronic Hospital Information System (HIS), contact with the general practitioner, referring cardiologist or the treating hospital. Cardiac death and nonfatal myocardial infarction are registered as major cardiac events. Cardiac death is defined as death from any cardiac cause (lethal arrhythmia, myocardial infarction, or congestive heart failure) or sudden unexpected death occurring without another explanation. Myocardial infarction is defined by angina of >30 minutes duration and either ST segment elevation of ≥2mm in 2 consecutive ECG leads or a rise in troponin T of ≥0.03µg/l.

Other events include clinically indicated coronary arterial revascularization by percutaneous coronary angioplasty (PCI) or coronary artery bypass graft (CABG).

In case of 2 simultaneous cardiac events, the worst event was selected (cardiac death>non-fatal myocardial infarction>revascularization).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before the MR-examination

Exclusion Criteria:

* Non-sinus rhythm, unstable angina, severe arterial hypertension (>200/120 mmHg), moderate or severe valvular disease and general contraindications to MRI (implanted pacemakers or defibrillators, intracranial metal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to our institution for clinically indicated dobutamine stress MRI due to suspected or known CAD (with/without prior revascularization and with/without history of previous myocardial infarction).
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2005-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cardiac death and nonfatal myocardial infarction (MACEs) | 2-5 years of follow-up

SECONDARY OUTCOMES:
Late revascularization (90 days after the MR-examination) | 2-5 yrs.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Department of Cardiology, Heidelberg, Germany

REFERENCES:
- [Derived] Korosoglou G, Elhmidi Y, Steen H, Schellberg D, Riedle N, Ahrens J, Lehrke S, Merten C, Lossnitzer D, Radeleff J, Zugck C, Giannitsis E, Katus HA. Prognostic value of high-dose dobutamine stress magnetic resonance imaging in 1,493 consecutive patients: assessment of myocardial wall motion and perfusion. J Am Coll Cardiol. 2010 Oct 5;56(15):1225-34. doi: 10.1016/j.jacc.2010.06.020. PMID 20883929